CLINICAL TRIAL: NCT04676568
Title: A One Year Interventional Study in Patients With Vesicovaginal Fistula
Brief Title: Comparative Analysis of Outcome Between Extravesical and Transvesical Repair for Vesico-vaginal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Urology, Rawalpindi (Other)
Responsible Party: Principal Investigator, Adnan Ali, Consultant Surgeon, Armed Forces Institute of Urology, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFIU
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Vesico Vaginal Fistula
MeSH Terms: conditions — Vesicovaginal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extravesical VVF repair (Active Comparator)
  Interventions: Procedure: Extravesical VVF repair
- Transvesical VVF repair (Active Comparator)
  Interventions: Procedure: Extravesical VVF repair

INTERVENTIONS:
Procedure: Extravesical VVF repair — Both standard transvesical and extravesical approach for VVF repair will be utilised
  Other Names: Transvesical VVF repair

SUMMARY:
In patients with vesicovaginal fistula, transvesical and extravesical repair will be compared in terms of operative time, complications and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* all patients with Vesicovaginal fistula

Exclusion Criteria:

* uretrovaginal fistula

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
operative time | 3 months
  total time taken for surgery
complications | 3 months
  bladder spasms, bleeding
recurrence | 3 months
  patients who have recurrenec of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of Urology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No